CLINICAL TRIAL: NCT04979169
Title: Increasing Lung Cancer Screening Uptake Among Emergency Department Patients
Brief Title: Emergency Department Lung Cancer URMFG Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, David Adler, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00006395
Record Dates: First submitted 2021-07-16; First posted 2021-07-28 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: The proposed study will utilize a randomized, prospectively collected, convenience sample and a longitudinal design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-adherent control (No Intervention): Subjects who are determined to be non-adherent to screening guidelines and are assigned to usual treatment via randomization in REDCap.
- Non-adherent intervention (Experimental): Subjects who are determined to be non-adherent to screening guidelines and are assigned to intervention treatment (text messaging) via randomization in REDCap.
  Interventions: Behavioral: Text Messaging

INTERVENTIONS:
Behavioral: Text Messaging — A series of theory-informed text messages encouraging them to contact their primary care provider and the UR LCS Program's Patient Navigator to coordinate screening, along with contact information to do so.
  Arms: Non-adherent intervention

SUMMARY:
This is a randomized controlled pilot trial of a text-based behavioral intervention aimed at increasing uptake of lung cancer screening among emergency department patients. We will conduct a 2-year randomized controlled clinical trial with a prospectively collected convenience sample of 366 adults who are eligible for LCS but non-adherent with LCS screening guidelines. Adults aged 50-80 will be recruited from a high-volume urban ED and a low-volume rural ED, assigned to study conditions, and followed-up at 150 days to assess interval engagement with the University of Rochester Medical Center's LCS screening program (primary outcome). Electronic Health Record (EHR) review will be conducted to assess screening results and subsequent clinical endpoints.

DETAILED DESCRIPTION:
Lung cancer is the number one cancer cause of death in the US1 accounting for a quarter of all cancer deaths. Five-year survival for lung cancer is just 19%. However, early detection of lung cancer increases 5-year survival three-fold and lung cancer screening (LCS) among high-risk patients using low-dose CT scan is cost-effective and has been proven to reduce lung cancer mortality by approximately 20%. Despite this potential, uptake of LCS has been poor with only 14.4% of eligible patients found to have been screened in a recent 10 state study. Indeed, the US Department of Health & Human Services and the USPSTF have both explicitly prioritized increasing the uptake of LCS among their goals. In 2021, the USPSTF revised the eligibility criteria for LCS, expanding the age range to 50-80 and lowering the pack-year threshold to 20.

The Emergency Department (ED) is an ideal setting to target an intervention aimed at increasing LCS uptake because the patient populations most in need are available for intervention. Our team has been at the forefront of ED-based cancer prevention efforts, serving as investigators on preventive work on cervical cancer and smoking cessation. EDs care for a disproportionate number of patients with the socio-economic factors that are associated with vulnerability to non-adherence with LCS including non-White race, lower income, and lack of health insurance. Moreover, smoking accounts for 90% of all lung cancer and ED patients have a higher smoking prevalence than the general population. In addition, ED visits generally involve periods of waiting during which preventive health needs can be assessed and intervened upon. LCS is a complex process - it is more than just an imaging study. However, the first critical step is to engage high-risk patients with this process. USPSTF has emphasized the importance of "pathways besides referral from primary care" to the success of this effort.

The vast majority of Americans - 95% - own a cell phone and an estimated 98% of all cell phones have SMS capabilities. Importantly, while there still exists a "digital divide" with regards to home computing among Americans of different backgrounds, phone ownership is nearly identical among white, black, and Hispanic Americans. SMS health interventions have been studied for over a decade and have been proven effective for a wide range of applications including smoking cessation, diabetes self care, and breast cancer screening. SMS interventions are low-cost, not staff-intensive, simple, familiar, scalable, tailorable to individuals, instantaneous in delivery, asynchronous in receipt, reproducible, and accessible regardless of geographical or socioeconomic factors. Our project adapts and targets this effective technology to improve LCS uptake among ED patients.

An empirically supported theoretical framework is central to developing an effective behavioral intervention, particularly in a setting like the ED where a long-term therapeutic relationship cannot be leveraged. The proposed trial makes use of two complementary theories: the Theory of Planned Behavior (TPB) and Self-Determination Theory (SDT). The TPB posits that the strongest predictor of a behavior is the intention to engage in the behavior. These intentions are predicted by an individual's attitudes toward the behavior, subjective normative beliefs about the behavior, and perceived control over whether they can perform the behavior. SDT states that individuals are motivated to engage in behaviors that satisfy the needs for (a) autonomy, (b) competence, and (c) relatedness. Individuals are autonomously motivated when these needs are met, which leads to engagement in a behavior.

The proposed study will utilize a randomized, prospectively collected, convenience sample and a longitudinal design with a sample size of 366 recruited from urban and rural UR Medicine EDs. Research enrollers will determine adherence of patients to USPSTF LCS recommendations using an adaptive REDCap survey. Non-adherent patients will be randomized to intervention or control conditions, with patients in the intervention condition receiving a series of theory-informed text messages encouraging them to contact their primary care provider and the UR LCS Program's Patient Navigator to coordinate screening, along with contact information to do so. Follow-up to determine LCS program uptake (primary outcome) will occur at 150 days, at which time feedback will also be solicited.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 - 80
* 20+ pack-year smoking history
* current smoker or quit within 15 years
* English, ASL, or Spanish speaking
* Presenting as a patient at the Strong Memorial or Noyes Community Hospital EDs

Exclusion Criteria:

* Non-English, Non-Spanish, and Non-ASL speaking
* Inability to consent (e.g. high clinical acuity)
* Lack of text-capable mobile phone and/or inability to use text function

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2021-12-08 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
Screening Uptake | 150 days
  Comparison of non-adherent intervention and control subjects for who are compliant with screening guidelines by the 150 day assessment

SECONDARY OUTCOMES:
Quality Indicators | 150 days
  Preliminarily assess quality indicators driven by engagement of study participants with the LCS program.
Barriers and Perceptions about Lung Cancer Screening | 150 days
  Qualitative analysis of subject feedback on barriers to obtaining screening and perceptions of the intervention in order to inform refinement and implementation of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: David Adler, MD, Principal Investigator — University of Rochester
Locations (1):
- Strong Hospital, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No